CLINICAL TRIAL: NCT00921622
Title: Vitamin Deficiency and Blood Pressure in Hospitalized JGH Patients
Brief Title: Vitamin Deficiency and Blood Pressure in Hospitalized Jewish General Hospital (JGH) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, John Hoffer, Physician, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-041
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Vitamin C Deficiency; Vitamin D Deficiency
Keywords: Blood pressure; Vitamin C; Vitamin D
MeSH Terms: conditions — Ascorbic Acid Deficiency; Vitamin D Deficiency | interventions — Vitamin D; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: vitamin C compared with vitamin D in prospective clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Active Comparator): 1000 IU twice daily for up to 10 days
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Vitamin C
- Vitamin C (Active Comparator): 500 mg twice daily for up to 10 days
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin D — 1000 IU twice daily for up to 10 days
  Arms: Vitamin D
Dietary Supplement: Vitamin C — 500 mg twice daily for up to 10 days

SUMMARY:
There is suggestive evidence that vitamin C and vitamin D deficiency may increase blood pressure across the range of blood pressures from normal to elevated. Information about this relationship is inadequate in part because of the rarity of individuals with subclinical vitamin C and D deficiency. The investigators have observed subnormal to deficient plasma vitamin C and 25-hydroxyvitamin D levels in a large proportion of patients under active treatment in the investigators' hospital. The clinical implications of widespread hypovitaminosis C and D are unknown. In this randomized prospective comparison trial the investigators will measure vitamin levels and blood pressure in clinically stable acutely hospitalized patients with a wide range of diagnoses, and expected to remain in the hospital for at least 7 more days. The investigators will examine for an inverse relationship between baseline vitamin level and blood pressure across the range of blood pressures. Consenting patients will be randomized to receive vitamin C (500 mg twice daily) or vitamin D (1000 IU twice daily) for as long as 10 days. Blood pressure will be re-measured every 2 days and vitamin levels re-measured on the last study day. Treatment courses of at least 5 days will be considered sufficient for analysis. The hypothesis is that either treatment will reduce blood pressure in patients whose baseline systolic blood pressure is 110 or more; the investigators will also examine whether the reduction in blood pressure with treatment is proportional to the increase in the circulating vitamin level with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Competent to grant informed consent
* Anticipated to remain in hospital at least 7 days after enrollment

Exclusion Criteria:

* End-stage renal disease on renal replacement therapy
* Critical illness
* Judged unstable clinical status at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
blood pressure | every 2 days for up to 10 days

SECONDARY OUTCOMES:
plasma vitamin levels: monitoring variable | at beginning and end of treatment course

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan R, Eintracht S, Hoffer LJ. Vitamin C deficiency in a university teaching hospital. J Am Coll Nutr. 2008 Jun;27(3):428-33. doi: 10.1080/07315724.2008.10719721. PMID 18838532